CLINICAL TRIAL: NCT04924400
Title: Complete Health Improvement Program to Improve Glycemic Control and Reduce Cost of Care for Geisinger Health Plan Members With Type 2 Diabetes
Brief Title: Complete Health Improvement Program for Geisinger Health Plan Members With Type 2 Diabetes
Acronym: CHIP-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Morland (Other)
Responsible Party: Sponsor-Investigator, Thomas Morland, Sponsor-Investigator, Geisinger Clinic
Organization: Geisinger Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-0438
Record Dates: First submitted 2021-05-20; First posted 2021-06-14 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHIP Program (Active Comparator): GHP members randomized to the intervention arm will participate in the CHIP Program.
  Interventions: Behavioral: CHIP Program
- Usual Diabetes Care (Active Comparator): GHP members assigned to the control arm will receive the routine standard of care for GHP members.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: CHIP Program — GHP members randomized to the intervention arm will participate in the following activities:
  * Attend 2 group meetings per week over 6 weeks, followed by one group meeting per week for 6 weeks (12 weeks total); each meeting will last about one hour. CHIP classes for weeks 1-4 and week 12 require in-person attendance, while week 5-11 classes can be attended either virtually or in-person.
  * Receive a copy of The Optimal Diet, The Official CHIP Cookbook.
  The following data will be collected at weeks 1,12 and 26:
  * Biometrics: weight, BMI, waist circumference, systolic and diastolic blood pressure
  * Biomarkers (blood tests): HbA1c, LDL-C
  * Psychometrics: Wellbeing360 survey
  Arms: CHIP Program
Behavioral: Usual Care — GHP members assigned to the control arm will receive the routine standard of care for GHP members. Members will receive a summary of diabetes-related benefits available to members with type 2 diabetes.
  The following data will be collected at weeks 1,12 and 26:
  * Biometrics: Weight, BMI, waist circumference, systolic and diastolic blood pressure
  * Biomarkers (blood tests): HbA1c, LDL-C
  * Psychometrics: Wellbeing360 survey
  Arms: Usual Diabetes Care

SUMMARY:
The Complete Health Improvement Program (CHIP) is a lifestyle improvement program intended to prevent and/or manage cardiovascular disease, diabetes, and other health conditions. This is a pilot-scale randomized-controlled trial comparing the clinical, utilization, and financial outcomes of adult health plan members with type 2 diabetes mellitus (T2DM) offered CHIP versus those only offered standard health plan coverage. We hypothesize that Geisinger Health Plan (GHP) members with T2DM offered CHIP in addition to standard insurance coverage will have improvement in HbA1c and improvements in other biometrics, biomarkers, psychometrics and utilization/financial outcomes, including LDL-C, systolic blood pressure, body mass index, waist circumference, number of diabetes medications prescribed, Wellbeing360 survey, and total cost of healthcare.

DETAILED DESCRIPTION:
This is a pilot prospective randomized-controlled trial of 60 patients randomized to either the intervention group; in which patients enroll in the CHIP program, or the control group, in which patients follow their usual diabetes care. We hypothesize that Geisinger Health Plan members with T2DM offered CHIP in addition to standard insurance coverage will have improvement in HbA1c and improvements in other biometrics, biomarkers, psychometrics and utilization/financial outcomes, including LDL-C, systolic blood pressure, body mass index, waist circumference, number of diabetes medications prescribed, Wellbeing360 survey, and total cost of healthcare.

The intervention group will attend 18 classes covering topics such as diet, sleep, exercise instruction, stress management, and toxic substance avoidance. Biometrics (weight, BMI, waist circumference, systolic/diastolic blood pressure), biomarkers (HbA1c, LDL-C) and psychometrics (Wellbeing 360 survey) will be collected on all participants at baseline, 3-months and 6-months.

The CHIP curriculum will be administered during twice weekly 1-hour classes over a 6-week period, followed by weekly 1-hour classes for an additional 6 weeks. The protocol will begin with a 1-month in-person period, with participants subsequently offered the choice between in-person and online attendance for the remaining sessions.

The primary aim is to compare change in HbA1c, LDL-C, systolic blood pressure, body mass index, and waist circumference for GHP members offered CHIP versus members offered standard insurance coverage at 3- and 6-months.

Through this pilot study, we hope to gain insight into whether and how such an application of CHIP could be a cost-effective tool for health plans such as GHP to achieve clinical and financial goals for adult members with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Geisinger Health Plan member for a full year prior to enrollment in the study, with plans to remain covered for a full year after the first study visit
* HbA1c resulted within a year of enrollment in the study
* ≥ 18 years
* Current type 2 diabetes diagnosis
* Living in the five-county region served by the Miller Center (Lycoming, Montour, Northumberland, Snyder and Union) with the ability to arrange their own transportation to the Miller Center in Lewisburg at least 10 times in a 3-month period
* Access to computer, phone, or tablet with sufficient internet to complete program activities.

Exclusion Criteria:

* Presence of medical condition requiring specific diet (e.g., Celiac disease, phenylketonuria)
* Presence of medical condition contraindicating participation in CHIP, as determined by the Principal Investigator (e.g. cancer on active treatment)
* Pregnancy or plan to become pregnant within one year
* Inability to give informed consent due to mental or psychiatric impairment
* Participation in the Fresh Food Farmacy program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas B Morland, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were sent letters and/or electronic portal messages inviting them to participate. Research staff followed up with recruitment phone calls.
Pre-assignment Details: Participants were randomized to the intervention versus control arms after providing informed consent.
Groups:
- CHIP Program: GHP members randomized to the intervention arm will participate in the CHIP Program.
  CHIP Program: GHP members randomized to the intervention arm will participate in the following activities:
  * Attend 2 group meetings per week over 6 weeks, followed by one group meeting per week for 6 weeks (12 weeks total); each meeting will last about one hour. CHIP classes for weeks 1-4 and week 12 require in-person attendance, while week 5-11 classes can be attended either virtually or in-person.
  * Receive a copy of The Optimal Diet, The Official CHIP Cookbook.
  The following data will be collected at weeks 1,12 and 26:
  * Biometrics: weight, BMI, waist circumference, systolic and diastolic blood pressure
  * Biomarkers (blood tests): HbA1c, LDL-C
  * Psychometrics: Wellbeing360 survey
- Usual Diabetes Care: GHP members assigned to the control arm will receive the routine standard of care for GHP members.
  Usual Care: GHP members assigned to the control arm will receive the routine standard of care for GHP members. Members will receive a summary of diabetes-related benefits available to members with type 2 diabetes.
  The following data will be collected at weeks 1,12 and 26:
  * Biometrics: Weight, BMI, waist circumference, systolic and diastolic blood pressure
  * Biomarkers (blood tests): HbA1c, LDL-C
  * Psychometrics: Wellbeing360 survey
Period: Overall Study
Arm/Group | CHIP Program | Usual Diabetes Care
Started (Please note discrepancy between overall number of patients enrolled and number listed participating. This is due to a flaw in the study design, in which patients underwent informed consent online from home, immediately after which randomization occurred. 38 participants provided informed consent and were randomized (19 participants to each arm), but 6 and 7 intervention and control participants, respectively) did not participate in any study activities following enrollment and randomization.) | 13 | 12 (Please note discrepancy between overall number of patients enrolled and number listed participating. This is due to a flaw in the study design, in which patients underwent informed consent online from home, immediately after which randomization occurred. 38 participants provided informed consent and were randomized (19 participants to each arm), but 6 and 7 intervention and control participants, respectively) did not participate in any study activities following enrollment and randomization.)
Completed | 10 | 12
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Population: 7 patients randomized to the control group did not attend baseline biomarkers/biometrics; 6 patients in the intervention group did not attend baseline biomarker/biometrics
Groups:
- Total: Total of all reporting groups
Arm/Group | CHIP Program | Usual Diabetes Care | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 7 | 19
  >=65 years | 1 | 5 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (9.27) | 60.9 (12.40) | 57.6 (11.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 11 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c
Description: Change in HbA1c after 6 months compared to baseline
Time Frame: 6 months
Population: Thirty-eight individuals consented to participated in this study. Nineteen were randomized to both the control and intervention groups. Seven intervention and eight control participants provided 6-month biomarkers/biometrics.
Measure: Mean (95% Confidence Interval); unit: Percentage of HbA1c
Arm/Group | CHIP Program | Usual Diabetes Care
Number analyzed (Participants) | 7 | 8
Percentage of HbA1c | -0.46 [-0.93 to -0.01] | -0.58 [-0.95 to -0.22]

2. Primary Outcome: Percentage of Patients Who Completed Biomarkers
Description: What percentage of individuals completed biomarkers
Time Frame: 3 and 6 months
Population: Thirty-eight individuals consented to participate in this study and 19 were randomized to both the control and intervention groups.
Measure: Count of Participants; unit: Participants
Arm/Group | CHIP Program | Usual Diabetes Care
Number analyzed (Participants) | 19 | 19
Participants
  Consented to participate but did not attend baseline biomarkers | 6 | 7
  Provided baseline biomarkers but no further biomarkers | 3 | 0
  Provided baseline and 3 month biomarkers only | 2 | 0
  Provided all biomarkers (baseline, 3-month, 6-month) | 8 | 12

3. Primary Outcome: Percentage of Patients Who Completed Biometrics
Description: What percentage of individuals completed biometrics
Time Frame: 3 and 6 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | CHIP Program | Usual Diabetes Care
Number analyzed (Participants) | 19 | 19
Participants
  Consented to participate but did not provide baseline biometrics | 6 | 7
  Provided baseline biometrics but no further biometrics | 3 | 0
  Provided baseline and 3 month biometrics only | 3 | 0
  Provided all biometrics (baseline, 3-month, 6-month) | 7 | 12

4. Primary Outcome: Percentage of Patients Contacted Who Agreed to Participate
Description: What percentage of individuals contacted who agreed to participate in the study
Time Frame: Baseline
Population: A total of 1,644 members were identified for recruitment and a letter was mailed to this group introducing the study. Of those who received a recruitment mailing, 1,087 members received at least one phone call to assess interest in participating in this study.
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Participants: GHP members meeting criteria for enrollment based upon electronic query of database available for preparation to research process. Members were contacted by letter, electronic portal, and/or telephone call. Participation rates are based upon patients excluded based upon inclusion/exclusion criteria, those who chose not to participate due to transportation issues, those who chose not to participate for another reason, and those who did consent to participate.
Arm/Group | Eligible Participants
Number analyzed (Participants) | 1644
Participants
  Members called at least once | 1087
  Unable to reach: number analyzed (Participants) | 1087
  Unable to reach | 690
  Did not meet inclusion/exclusion criteria after telephone screening: number analyzed (Participants) | 1087
  Did not meet inclusion/exclusion criteria after telephone screening | 8
  Declined due to transportation issues: number analyzed (Participants) | 1087
  Declined due to transportation issues | 53
  Declined for another reason: number analyzed (Participants) | 1087
  Declined for another reason | 254
  Consented to participate in the study: number analyzed (Participants) | 1087
  Consented to participate in the study | 38

5. Secondary Outcome: HbA1c Control at 3 Months
Description: Change in HbA1c percentage at 3 months compared to at baseline
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: Percent
Arm/Group | CHIP Program | Usual Diabetes Care
Number analyzed (Participants) | 10 | 12
Percent | -0.92 [-1.81 to -0.03] | -0.58 [-0.95 to -0.22]

6. Secondary Outcome: LDL-C at 3 Months
Description: Change in LDL-C levels at 3 compared to baseline
Time Frame: 3 months
Population: Nineteen individuals were randomized to each group. Some participants did not return for the 3 and/or 6 month biomarker/biometric collection, resulting in fewer participants being included in the analysis at these timepoints.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | CHIP Program | Usual Diabetes Care
Number analyzed (Participants) | 10 | 12
mg/dL | -4.11 [-15.48 to 7.25] | -8.58 [-25.80 to 8.63]

7. Secondary Outcome: Change in Weight at 3 Months
Description: Change in weight at 3 months compared to baseline
Time Frame: 3months
Measure: Mean (95% Confidence Interval); unit: Pounds
Arm/Group | CHIP Program | Usual Diabetes Care
Number analyzed (Participants) | 9 | 12
Pounds | -5.15 [-11.02 to 0.72] | -2.22 [-4.86 to 0.42]

8. Secondary Outcome: Change in Weight at 6 Months
Description: Change in weight at 6 months compared to baseline
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: Pounds
Arm/Group | CHIP Program | Usual Diabetes Care
Number analyzed (Participants) | 7 | 12
Pounds | -7.38 [-15.49 to 0.74] | -2.10 [-5.69 to 1.49]

9. Secondary Outcome: Health Behaviors, as Measured by CHIP Participation
Description: Overall program completion, defined as completing the majority of study activities
Time Frame: 6 months
Population: Participation in at least half of designated study activities
Measure: Count of Participants; unit: Participants
Arm/Group | CHIP Program | Usual Diabetes Care
Number analyzed (Participants) | 13 | 12
Participants | 9 | 12

10. Secondary Outcome: Number of Diabetes Medications Prescribed at 6 Months
Description: Change in number of diabetes medications at 6 months compared to baseline. Number of diabetes medications, by medication class, were collected for each responding patient at 3 and 6 months. Due to small sample size and lack of reversing changes between 3 and 6 months (i.e. all changes made by 3 months were continued at 6-month mark, whereas some additional changes were made between 3 and 6 months), changes between months 1-3 and 4-6 were pooled into a single report of cumulative change between baseline and the 6-month mark).
Time Frame: 6 months
Measure: Mean (Full Range); unit: Medications
Arm/Group | CHIP Program | Usual Diabetes Care
Number analyzed (Participants) | 9 | 12
Medications | -0.11 [-1 to 1] | 0.50 [-1 to 1]

11. Secondary Outcome: Change in LDL-C at 6 Months
Description: Change in LDL-C at 6 months compared to baseline
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | CHIP Program | Usual Diabetes Care
Number analyzed (Participants) | 8 | 12
mg/dL | -4.71 [-20.30 to 10.87] | -8.58 [-25.80 to 8.63]

12. Secondary Outcome: Systolic Blood Pressure After 3 Months
Description: Change in systolic blood pressure at 3 months compared to baseline
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | CHIP Program | Usual Diabetes Care
Number analyzed (Participants) | 9 | 12
mm Hg | -4.50 [-12.54 to 3.54] | -16.00 [-26.02 to -5.98]

13. Secondary Outcome: Systolic Blood Pressure at 6 Months
Description: Change in systolic blood pressure at 6 months compared to baseline
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | CHIP Program | Usual Diabetes Care
Number analyzed (Participants) | 7 | 12
mm Hg | 4.13 [-8.89 to 17.14] | -4.83 [-14.46 to 4.79]

14. Secondary Outcome: Diastolic Blood Pressure at 6 Months
Description: Change in diastolic blood pressure at 6 months compared to baseline
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | CHIP Program | Usual Diabetes Care
Number analyzed (Participants) | 7 | 12
mm Hg | 1.13 [-4.93 to 7.18] | -1.00 [-5.68 to 3.68]

15. Secondary Outcome: Diastolic Blood Pressure After 3 Months
Description: Change in diastolic blood pressure at 3 months compared to baseline
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | CHIP Program | Usual Diabetes Care
Number analyzed (Participants) | 9 | 12
mm Hg | 0.40 [-4.36 to 5.16] | -4.83 [-11.57 to 1.90]

16. Secondary Outcome: Change in Total Cost of Care, Versus Same 6 Months Year Prior
Description: This outcome evaluates cost of care in the 6 months beginning to the first day of the CHIP program versus the same 6 months as patient's participation in the study one year prior to enrollment
Time Frame: 6 months of participation compared to same period one year prior
Population: Please note discrepancy between number of patients analyzed and those enrolled/randomized. Individuals randomized to either the intervention or control who completed to study activities (i.e. did not attend any biomarker/biometric collections or CHIP classes) were excluded. Participants in the intervention and control group who gave baseline biomarkers and/or biometrics were included in the cost analyses
Measure: Mean (Standard Deviation); unit: Dollars
Units Other Than Participants: dollars
Arm/Group | CHIP Program | Usual Diabetes Care
Number analyzed (Participants) | 13 | 12
Number analyzed (dollars) | 1 | 1
Dollars | -859 (12161) | 1303 (2870)

17. Secondary Outcome: Change in Total Cost of Care Versus 6 Months Leading to Intervention
Description: This outcome evaluates cost of care in the 6 months beginning to the first day of the CHIP program versus the 6 months leading up to that date
Time Frame: 6 months beginning with first day of intervention versus 6 months leading up to that day
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | CHIP Program | Usual Diabetes Care
Number analyzed (Participants) | 13 | 12
Dollars | 1174 (5001) | -97 (1628)

ADVERSE EVENTS:
Time Frame: Adverse events were not tracked for this minimal risk study.
Description: There was not formal monitoring for Serious Adverse Events. The study team is not aware of any deaths or serious adverse events among intervention or control participants.
Arm/Group | Usual Diabetes Care
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
This was a pilot and feasibility study, not powered to answer questions regarding the effect of the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/00/NCT04924400/Prot_SAP_000.pdf